CLINICAL TRIAL: NCT01795677
Title: JAK2 Inhibitors RUXOLITINIB in Patients With High or Intermediate Risk Primary or Secondary Myelofibrosis Eligible for Allogeneic Stem Cell Transplantation: a Prospective Multicentric Phase II Study
Brief Title: JAK2 Inhibitors RUXOLITINIB in Patients With Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JAK ALLO STUDY
Record Dates: First submitted 2012-12-21; First posted 2013-02-21 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Myelofibrosis
Keywords: JAK2 inhibitor RUXOLITINIB; Primary or secondary myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RUXOLOTINIB (Experimental): Ruxolotinib : patient with donor HSCT 4 months later patients without donor: ruxolotinib alone
  Interventions: Drug: Ruxolotinib

INTERVENTIONS:
Drug: Ruxolotinib — Ruxolotinib doses calculated with platelets count and P450 cytochrome inhibitor HSCT for patients with donor
  Other Names: Kakavi

SUMMARY:
JAK2 inhibitor RUXOLITINIB before allogeneic hematopoietic stem cell transplantation (HSCT) in patients with primary or secondary myelofibrosis : a prospective phase II

DETAILED DESCRIPTION:
JAK2 inhibitor RUXOLITINIB before allogeneic hematopoietic stem cell transplantation (HSCT) in patients with primary or secondary myelofibrosis

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 69 years
* No comorbidity contraindicating the transplantation :

  * Severe respiratory failure defined as dyspnea grade III or more
  * Severe cardiac failure defined as EF < or = 30%
  * Severe renal failure defined as creatinine clearance < 30 ml/min or dialysis
  * Dementia or non-ability to give informed consent for the protocol
  * Major alteration of performance status defined as ECOG > 2
  * Severe liver disease defined as a cirrhosis or bilirubin > 2 x ULN, or AST/ALT > 5 x ULN
* Primary or secondary myelofibrosis diagnosed according to WHO definition (Tefferi, et al 2007)
* Palpable splenomegaly or splenomegaly measured by any imagery (maximum size> 15 cm by ultrasound scan, Magnetic Resonance Imaging or computer tomography)
* Disease if intermediate or high risk according to published criteria and summarized as follows:

At least one criterion among the following:

* Haemoglobin < 100 gr/L (unrelated to medication toxicity)
* Leucocytes < 4 G/L (unrelated to medication toxicity) or > 25 G/L
* Poor prognosis cytogenetics : complex karyotype, abnormalities of chromosomes 5, 7 or 17 , +8, 12p-, inv(3), 11q23

Two criteria among the following criteria :

* General symptoms (weight lost > 10% in less than 6 months, night swears, specific fever > 37.5°C)
* Peripheral blastosis > 1% observed at least twice
* Thrombocytopenia < 100 G/L (unrelated to treatment toxicity)

Exclusion Criteria:

* Myelofibrosis transformed into acute leukaemia with 20% blasts of more in blood or bone marrow
* Previous treatment with JAK2 inhibitor
* Thrombopenia < 50 G/L
* Comorbidities contraindicating the transplantation
* Comorbidity score Sorror > 3
* Pregnant or lactating women

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-12; Primary Completion 2018-05 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
DFS | 24 months after inclusion
  DFS is defined as the probability to be alive and in remission

SECONDARY OUTCOMES:
HSCT | 24 months after inclusion
  * Rate of pre-graft splenectomy
  * Co-morbidity score defined by Sorror et al before RUXOLITINIB and after 4-month treatment just before transplantation
  * Post-graft haematological recovery: time to neutrophil engraftment, platelet and red blood cells transfusion independency
  * Acute GVHD grade II-IV incidence
  * Chronic GVHD incidence
  * Overall survival, disease-free survival, non-relapse mortality
  * JAK2V617E allele burden and status at registration, 3, 7, 16 months after inclusion (centralization)
PATIENTS CARACTERISTICS | 24 months after inclusion
  Patients with and without donor
  * Rate of patients with donor who benefit from a transplantation:
  * Comorbidity score at registration and after 3 months
  * Platelet and red blood cells transfusion independency
  * Performance status evolution (ECOG)
  * General symptoms related to myelofibrosis (questionnaire MF SAF)
  * Comparison of haematological response in patients with or without donor
  * Spleen size evolution
  * Comparison of quality of life in patients with and without (questionnaire EORTC)
  * Comparison of overall survival in patients with and without donor
  * Incidence of severe infections
  * Cytokine measure at registration, 3, and 7 months after inclusion (centralization)
  * MPL JAK status (at registration, centralization

CONTACTS AND LOCATIONS:
Overall Officials: MARIE ROBIN, MD, Principal Investigator — FIM/GOELAMS
Locations (1):
- ROBIN, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FILO internet site — http://www.filo-leucemie.org